CLINICAL TRIAL: NCT04784702
Title: Smoking Cessation in Patients After Coronary Angiography - Self-achieved and Supported With Cytisine and Its' Effect on Platelet Aggregation
Brief Title: Smoking Cessation in Patients After Coronary Angiography
Status: Completed | Type: Observational
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Bogumil Ramotowski, MD, PhD, Adjunct, Director of the Programme, Centre of Postgraduate Medical Education
Other Study IDs: 16/PB/2014
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
OBJECTIVES The goal of this study is to evaluate the self-achieved smoking cessation supported with cytisine smoking cessation and its' on platelet aggregation and prothrombotic state in patients after coronary angiography and PCI.

BACKGROUND Cigarette smoking is a major risk factor of coronary artery disease (CAD). Smoking cessation is one of the most cost-effective intervention in lifestyle. Self-reported rates of smoking cessation are reasonably low. Cytisine is promising drug in support of smoking cessation. Smoking affects various components leading to arterial thrombosis, and the effect of smoking cessation on prothrombotic state and platelet aggregation is still under investigation GOAL To assess rates of smoking cessation in patients after coronary angiography and PCI and factors influencing success in smoking cessation To assess feasibility, safety and efficacy of cytisine in smoking patients To assess effect of smoking cessation on platelet aggregation in patients treated with clopidogrel and on prothrombotic state.

METHODS A prospective nonrandomized observational study of patients after coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients after coronary angiography or PCI,
* Aged 18 years or older,
* Smoking at least 10 cigarettes a day

Exclusion Criteria:

• Pregnancy

Criteria may vary in substudies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable CAD and ACS admitted to the catheterization laboratory in the Department of Cardiology, Grochowski Hospital, Warsaw, Poland
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation in patient treated with clopidogrel after smoking cessation | 30-days
  Platelet reactivity measured with PRU

SECONDARY OUTCOMES:
Prothrombotic state | 30-days
  Various biomarkers
Cotinine | 30-days
  Changes in concentration of cotinine
Thrombin potential | 30-day
  Assessment of endogenous thrombin potential
Thrombomodulin | 30-days
  Changes of thrombomodulin concentration
PAI-1 | 30-days
  Changes of PAI-1 concentration
P-selectin | 30-days
  Changes of p-selectin concentration
PF-4 | 30-days
  Changes of PF-4 concentration
Thromboglobulin | 30-days
  Changes of thromboglobulin concentration

OTHER OUTCOMES:
Smoking cessation | 30-days, 6-months, 12-months
  Factors influencing smoking cessation. Smoking cessation assessed with NicAlert test and self-reported
Cytisine as smoking cessation aid | 30-days
  Feasibility,safety and effectiveness of cytisine. Number of patients with confirmed smoking cessation.Number of adverse events